CLINICAL TRIAL: NCT01026545
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of PF-04287881 After Administration Of Multiple Escalating Oral Doses To Healthy Adult Subjects
Brief Title: Multiple Oral Dose Safety, Tolerability And Pharmacokinetic Study Of PF-04287881 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B0581002
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Respiratory Tract Infections
Keywords: safety; tolerability; pharmacokinetics; multiple-dose; macrolide
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 2 (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 3 (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 4 (optional) (Experimental): If intermediate or repeat dose level is needed; dose will not exceed 1100 mg.
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 5 (Japanese) (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 6 (Japanese) (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo

INTERVENTIONS:
Drug: PF-04287881 — 500 mg once daily for 10 days
  Arms: Cohort 1
Drug: Placebo — To match 500 mg dose once daily for 10 days
  Arms: Cohort 1
Drug: PF-04287881 — 750 mg once daily for 10 days
  Arms: Cohort 2
Drug: Placebo — To match 750 mg dose once daily for 10 days
  Arms: Cohort 2
Drug: PF-04287881 — 1100 mg once daily for 10 days
  Arms: Cohort 3
Drug: Placebo — To match 1100 mg dose once daily for 10 days
  Arms: Cohort 3
Drug: PF-04287881 — Optional cohort with dose not greater than 1100 mg
  Arms: Cohort 4 (optional)
Drug: Placebo — Optional cohort to match dose not greater than 1100 mg
  Arms: Cohort 4 (optional)
Drug: PF-04287881 — 750 mg dose once daily for 10 days
  Arms: Cohort 5 (Japanese)
Drug: Placebo — To match 750 mg dose once daily for 10 days
  Arms: Cohort 5 (Japanese)
Drug: PF-04287881 — 1100 mg dose once daily for 10 days
  Arms: Cohort 6 (Japanese)
Drug: Placebo — To match 1100 mg dose once daily for 10 days
  Arms: Cohort 6 (Japanese)

SUMMARY:
This study is a randomized, investigator blind, subject blind, sponsor-open, placebo controlled, multiple dose escalating, sequential, parallel cohort study of PF-04287881. Subjects will undergo screening procedures within 28 days prior to dosing. At least 1 day after the Screening visit, eligible subjects who meet the entry criteria will be admitted to the Clinical Research Unit (CRU) and confined in the unit until discharge on Day 15.

Approximately 60 healthy volunteers (20 volunteers of Japanese origin for Cohorts 5 and 6), 18 to 55 years of age, males and females (women of non childbearing potential only) will be enrolled and randomized in a 4:1 ratio to treatment with either PF-04287881 or placebo within each cohort. Each cohort will have a 10 day dosing period and each will consist of 10 subjects (8 active and 2 placebo). In each cohort, each subject will receive a single daily oral dose of either placebo or PF-04287881 under fasted state for 10 days.

DETAILED DESCRIPTION:
Following a Serious Adverse Event (potential Hy's Law case), a risk-benefit assessment review of all preliminary safety data, and a review by Pfizer's internal hepatic injury advisory panel, it was concluded that PF-04287881 had an unacceptable therapeutic window. The FDA was notified of our intention to discontinue development as of 09April2010.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers willing and able to be confined to the Clinical Research Unit and comply with study schedule.
* Women of non-childbearing potential only.
* Japanese subjects must have 4 Japanese grandparents who were born in Japan.

Exclusion Criteria:

* Previous antibiotic use within 14 days prior to dosing.
* Use of antibiotics during hospitalization within 90 days prior to dosing.
* History of hypersensitivity to macrolides or ketolides.
* Presence of clinically significant eye conditions (other than corrective lenses).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Standard safety assessments including assessment of AEs, laboratory tests, ECGs, and vital signs. | Screening, Dosing days 1-10, through follow-up
The primary pharmacokinetic endpoints to be evaluated for PF-04287881 include Cmax, Tmax, and AUC(0-24) on Day 1 and Day 10. | Day 1 and 10

SECONDARY OUTCOMES:
Secondary parameters include AUCinf and t1/2 as data permit, apparent oral clearance (CL/F), apparent volume of distribution (Vz/F) and accumulation ratio (Rac). | Days 1, 5 and 10
Urine concentrations of PF 04287881 in Cohorts 2 and 5 will be used to determine total amount excreted (Ae), %Ae relative to dose given and renal clearance (CLR). | Day 10
Concentrations of PF 04287881 will be measured in white blood cell (WBC) polymorphonuclear cells (PMNs) in Cohorts 2 and 5 to determine total exposure in WBC. | Days 1 and 10
Plasma samples from Cohort 2 will be used for exploratory investigation of circulating metabolites. | Days 1 and 10

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0581002&StudyName=Multiple%20Oral%20Dose%20Safety%2C%20Tolerability%20And%20Pharmacokinetic%20Study%20Of%20PF-04287881%20In%20Healthy%20Adult%20Subjects